CLINICAL TRIAL: NCT06032923
Title: Double-blind Placebo Controlled Study to Evaluate the Effect of NAD+ Boosting With Nicotinamide Riboside on Immunometabolism and Immunity in Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10001621; 001621-H
Record Dates: First submitted 2023-09-09; First posted 2023-09-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06-05

CONDITIONS: Systemic Lupus Erythematosus (Sle)
Keywords: Lupus; Chronic Inflammation
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy controls (No Intervention): This group will not receive the dietary supplement or placebo.
- Subjects with SLE - Active (Active Comparator): This study group will take the dietary supplement Nicotinamide Riboside capsules.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Subjects with SLE - Placebo (Placebo Comparator): This study group will take the Placebo.
  Interventions: Dietary Supplement: Nicotinamide Riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — The dietary supplement Nicotinamide Riboside or a placebo capsule in subjects with SLE. Niagen(R) is a commercially available form of nicotinamide riboside (NR)
  Arms: Subjects with SLE - Active; Subjects with SLE - Placebo

SUMMARY:
Study Description:

Systemic lupus erythematosus (SLE) occurs predominantly in women and is driven by type I interferon dysregulation and neutrophil hyperresponsiveness. Neutrophils in females have reduced mitochondrial bioenergetic capacity which affects immunometabolism. Nicotinamide adenine dinucleotide (NAD)+ boosting with nicotinamide riboside blunts type 1 IFN activation in-vivo in monocytes of healthy subjects and ex-vivo in SLE subjects. These findings support the proposal of the hypothesis that NAD+ boosting by NR supplementation will modulate metabolic pathways in lupus and blunt type 1 interferon signaling. Moreover, as type 1 interferon drives endothelial dysfunction, linked to increased cardiovascular risk, the effect of NR on endothelial function will be examined.

Objectives:

Primary Objective: Evaluate the effect of NR vs. placebo on immunometabolic and inflammatory remodeling in female SLE subjects:

Exploratory Objective: Compare and characterize myeloid cell bioenergetic and immunometabolic profiles in healthy control and SLE female subjects

Endpoints:

Primary Endpoint:

The primary end point will be to assess the effect of NR on blunting type I IFN signaling by measuring monocytic secretion of IFN-beta secretion compared to baseline in response to placebo vs. NR supplemented in SLE study subjects.

Exploratory Endpoints:

Healthy control vs. SLE subjects:

* Compare type I IFN transcript profiles in monocytes and neutrophils at baseline and in response to activation.
* Assess cell bioenergetics including: 1) monocyte and neutrophil metabolic flux mass spectroscopy of 13C-glucose and 13Cglutamine analysis to investigate their metabolic fates; (iii) Mitochondrial oxygen consumption (using glucose, amino acid, and fatty acid substrates) and glycolysis rates.

SLE baseline vs. NR/placebo supplementation:

Baseline vs. 6 weeks of NR/placebo:

-Assess effect of NR on bioenergetics by measuring steady-state metabolite levels comparing changes in placebo vs. NR groups in monocytes and neutrophils.

Baseline vs. 12 weeks of NR/placebo:

* Whole blood NAD+ levels (batched and measured at the end of study enrollment period)
* Explore effects of NR on gene regulation using monocyte and neutrophils by RNA-seq and chromatin remodeling analysis.
* Determine the effect of NR vs placebo on endothelial dysfunction in SLE subjects

DETAILED DESCRIPTION:
Study Description:

Systemic lupus erythematosus (SLE) occurs predominantly in women and is driven by type I interferon dysregulation and neutrophil hyper-responsiveness. Neutrophils in females have reduced mitochondrial bioenergetic capacity which affects immunometabolism. Nicotinamide adenine dinucleotide (NAD)+ boosting with nicotinamide riboside blunts type 1 IFN activation in-vivo in monocytes of healthy subjects and ex-vivo in SLE subjects. These findings support the proposal of the hypothesis that NAD+ boosting by NR supplementation will modulate metabolic pathways in lupus and blunt type 1 interferon signaling. Moreover, as type 1 interferon drives endothelial dysfunction, linked to increased cardiovascular risk, the effect of NR on endothelial function will be examined.

Objectives:

Primary Objective: Evaluate the effect of NR vs. placebo on immunometabolic and inflammatory remodeling in female SLE subjects:

Exploratory Objective: Compare and characterize myeloid cell bioenergetic and immunometabolic profiles in healthy control and SLE female subjects

Endpoints:

Primary Endpoint:

The primary end point will be to assess the effect of NR on blunting type I IFN signaling by measuring monocytic secretion of IFN-beta secretion compared to baseline in response to placebo vs. NR supplemented in SLE study subjects.

Exploratory Endpoints:

Healthy control vs. SLE subjects:

* Compare type I IFN transcript profiles in monocytes and neutrophils at baseline and in response to activation.
* Assess cell bioenergetics including: 1) monocyte and neutrophil metabolic flux mass spectroscopy of 13C-glucose and 13C-glutamine analysis to investigate their metabolic fates; (iii) Mitochondrial oxygen consumption (using glucose, amino acid, and fatty acid substrates) and glycolysis rates.

SLE baseline vs. NR/placebo supplementation:

Baseline vs. 6 weeks of NR/placebo:

-Assess effect of NR on bioenergetics by measuring steady-state metabolite levels comparing changes in placebo vs. NR groups in monocytes and neutrophils.

Baseline vs. 12 weeks of NR/placebo:

* Whole blood NAD+ levels (batched and measured at the end of study enrollment period)
* Explore effects of NR on gene regulation using monocyte and neutrophils by RNA-seq and chromatin remodeling analysis.
* Determine the effect of NR vs placebo on endothelial dysfunction in SLE subjects

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

SLE subjects:

* Female subjects 18 years or older who meets > 3 of 11 modified Am. Coll. of Rheumatology (ACR) (1997) Revised Criteria for SLE and mild/moderate disease activity defined as an SLE Disease Activity Index 2000(SLEDAI 2K) between zero and less than or equal to 14 at screening;
* If on glucocorticoids, the dose must be less than or equal to 20 mg daily and stable for at least 4 weeks prior to screening;
* If on hydroxychloroquine or other antimalarials such as chloroquine or quinacrine, dose must have been stable for the 12 weeks prior to screening. The max. allowed doses - hydroxychloroquine 400 mg/day, chloroquine phosphate 500 mg/day and quinacrine 100 mg/day;
* If on immunosuppressive drugs (methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus); dose must have been stable for the 12 weeks prior to screening
* Subjects of childbearing potential must agree to practice effective birth control for the duration of the study;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* Agreement to adhere to Lifestyle Considerations throughout study duration;
* Ability of subject to understand and the willingness to sign a written informed consent document.
* If on vitamin B3 or tryptophan supplementation at screening, willing to stop it at least 6 weeks before the baseline visit.

Control subjects:

* Female subjects 18 years or older
* No history of autoimmune or inflammatory disease
* If on vitamin B3 or tryptophan supplementation at screening, willing to stop it at least 6 weeks before the blood draw visit.

EXCLUSION CRITERIA:

SLE Subjects:

* Active renal or central nervous system disease or major renal or hepatic dysfunction;
* Treatment with rituximab, belimumab or any other biologic agent within the 6 months prior to screening
* Treatment with cyclophosphamide or IVIG within the 6 months prior to screening and or increase in glucocorticoid dose within 4 weeks of screening;
* Pregnancy or lactation (nursing)
* Treatment with another investigational drug or other intervention within 6 months of screening

Control Subjects:

* Inability to sign consent
* Pregnancy or nursing

Pregnant women are excluded from participation on this study. Self-reported pregnancy status may be accepted from female control participants of child-bearing potential for a blood draw which is considered a minimal risk procedure.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary end point will be to assess the effect of NR on blunting type I IFN signaling and cytokine secretion from placebo vs. NR supplemented subjects in monocytes comparing baseline (visit 1 to visit 3). | 4 years
  Type 1 IFN dysregulation is present in SLE. NAD+ boosting blunts type 1 interferon in healthy subjects in-vivo and in monocytes of SLE subjects ex-vivo. Completion of data collection time is by 01/2027.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001621-H.html